CLINICAL TRIAL: NCT05664282
Title: Orthodontic Treatment in Adolescents With Crowding and Displaced Teeth From the Clinical, the Patients' and Economic Perspectives
Brief Title: Orthodontic Treatment in Adolescents With Crowding and Displaced Teeth
Acronym: CROWDIT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Malmö University (Other)
Responsible Party: Principal Investigator, Liselotte Paulsson, Associate Professor, Malmö University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FO 2022/474
Record Dates: First submitted 2022-11-24; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Crowding, Tooth; Orthodontic
Keywords: tooth alignment; function; adverse side effects; cost-effectiveness
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Damon self-ligating brackets (Active Comparator): A multi-centre two-arm parallel-group randomized controlled trial with a 1:1 allocation ratio, comparing/evaluating tooth alignment, function and adverse side effects, Patients' perception of pain, function and quality of life Cost-effectiveness for adolescents with crowding and displaced teeth treated with self-ligating (Damon).
  Interventions: Device: Damon self-ligating brackets
- Victory conventional brackets (Active Comparator): A multi-centre two-arm parallel-group randomized controlled trial with a 1:1 allocation ratio, comparing/evaluating tooth alignment, function and adverse side effects, Patients' perception of pain, function and quality of life Cost-effectiveness for adolescents with crowding and displaced teeth treated with conventional brackets (Victory).
  Interventions: Device: Victory self-ligating brackets

INTERVENTIONS:
Device: Damon self-ligating brackets
  Arms: Damon self-ligating brackets
Device: Victory self-ligating brackets
  Arms: Victory conventional brackets

SUMMARY:
The purpose is to fill knowledge gaps identified for orthodontic treatment using a novel study design that has not been implemented in the dental field or in orthodontics. The study design comprises an analysis, where outcomes of two techniques are assessed at several efficacy levels by different methods. Moreover, the project is designed to include a longtime follow-up that is unique in orthodontic treatment. The aim is to compare two techniques with buccally fixed appliance in a multicenter RCT of adolescents aged 12 to 17 years with crowding and tooth displacement. In the intervention group, patients will be treated with a self-ligating bracket system, and in the control group with a conventional bracket system. Outcomes will be assessed from the clinical, patients' and economic perspectives as:

* Tooth alignment, function and adverse side effects
* Patients' perception of pain, function and quality of life
* Cost-effectiveness.

DETAILED DESCRIPTION:
Overall project design The primary outcomes of treatment will be tooth alignment and function on the clinical level. Other outcomes on the clinician's, patients and societal levels as well as adverse effects will be considered as secondary outcomes. The treatment consists of two phases, first an active treatment phase with fixed appliance during 2 years to align the arches. Secondly, the so called retention treatment, aimed at stabilization and maintenance of the achieved correction. This means that the active treatment and follow-up will last for 7 (2+5) years.

Subjects The patients, recruited from four orthodontic specialist clinics (two clinics in Region Skåne), are boys and girls aged 12 to 17 years with crowding and tooth displacement. Adolescents with craniofacial syndromes, previous orthodontic treatment, ongoing sucking habits and persisting primary teeth will be excluded as well as patients with crowding and displacement treated with extraction. The patients will be randomized in two groups and treated to a pre-set standard concept developed for each treatment group, the conventional with bracket system (Straight-wire, 3M®) and the new with self-ligating bracket system (Damon®). The randomization will follow recommendation from the CONSORT group. A statistician will perform the randomization for all clinics according to "Permuted block design" with equal number in both groups. To obtain the (random) sequence, a computerized random-number generator will be used.

Power analysis To test the null hypothesis that the two population means are equal on tooth alignment and function the criterion for significance (alpha) has been set at 0.050. The test is 2-tailed, i.e. an effect in either direction will be interpreted. With the proposed sample size of 75 in each group, the study will have power of 86% to yield a statistically significant result. The computation assumes that the mean difference is 500 SEK and the common within-group standard deviation is 1000 SEK. This was selected as the smallest effect that would be important to detect, in the sense that any smaller effect would not be of substantive significance.

Key action 1 - Evaluating the treatment methods at the clinicians' level Specific aim 1: To compare the techniques on ease of use, time at chairside and for maintenance Rationale: Orthodontic treatment with fixed appliance demands technical skill and is time-consuming. Therefore it is motivated to evaluate the techniques with regard to ease of use, time at chairside and time for maintenance. The new technique, self-ligating bracket system, is supposed to produce low-forces due to low-friction and this should facilitate more efficient tooth movement,extended intervals between appointments and reduction of chairside time. Presently there is insufficient evidence to support these assumptions. Methods: Protocols of the treatment with the techniques will be used to document treatment time, number of visits, defaults and cancellations. Expected outcome: We expect to find the self-ligating technique to result in shorter total treatment time compared with the conventional technique. The self-ligating technique will also be easier and quicker to handle when changing wires.

Key action 2 - Evaluating treatment outcomes at the clinical level Specific aim 2: To evaluate tooth alignment, function and morphological stability of the techniques under comparison Rationale: The goal of orthodontic treatment is to achieve an occlusion with good function, esthetical appearance and long- term stability. Immediately following completed treatment results are usually satisfactory with ideal occlusion and appearance. The few long-term studies indicate that during a follow-up time of at least 5 years crowding often arise.

Methods: Protocols will follow each patient throughout the treatment and follow-up. The patients will be documented with dental casts, photography and radiography at baseline, after 9-12 months treatment, at end of active treatment and at 7 years after treatment start. To evaluate tooth alignment, function stability and treatment success Little´s irregularity index (index to score mandibular incisor alignment) and Weighted Peer Assessment Rating index (PAR) will be used on dental casts. PAR scores are assigned to different malocclusion traits and the difference between pre- and posttreatment scores indicates the degree of improvement as a result of orthodontic intervention. Expected outcome: The techniques will result in equal results on tooth alignment and treatment success. The new technique is based on a different pattern of tooth movement and may result in a better long-term stability compared to the conventional technique.

Specific aim 3: To evaluate root resorption and marginal bone loss after treatment Rationale: Adverse side effects on hard tissues caused by orthodontic treatment, such as root resorption and loss of the marginal bone tissue, occur. As changes of the buccal and palatinal parts of roots and bone tissue are difficult to visualize by intraoral radiography, these side effects have been underestimated. CBCT that permits 3-D imaging has revealed that in patients treated with fixed appliances root resorption occurs in 94% of the patients and there are extensive changes of the marginal bone tissue lingually and buccally. The long-term analysis of these side effects comprises previously untouched terrain in research on orthodontic treatment. Methods: Clinical and radiographic examinations will be performed at baseline, after 9-12 months, at end of active treatment and at 5 years after treatment. Intraoral radiography and CBCT will be performed to examine the tooth roots and supporting bone tissue. To evaluate gingival recession study casts, intraoral photographs and probing depth will be used.

Expected outcome: The severity of changes will be smaller with the new technique as it is said to cause reduced frictional resistance and less forces. Root resorption and marginal bone loss will be more extensive than found previously in orthodontic treatment. Specific aim 4: To evaluate caries development Rationale: The scientific evidence is insufficient whether orthodontic treated patients develop more initial (white spot lesions) or manifest carious lesions compared to untreated indiviuals. Carious lesions may be underestimated and there is a lack of longterm analysis of these lesions. Methods: Clinical examination, bitewing radiographs and intraoral photographs will be performed at baseline, at end of active treatment and 7 years after treatment start to examine initial and manifest carious lesions at all tooth surfaces .

Expected outcome: We expect that carious increment will be less with the new technique due to less plaque accumulation and shorter treatment time. Key action 3 - Evaluating treatment outcomes on the patient's level Specific aim 5: To assess pain experienced by the patients Rationale: It is said that the lower orthodontic forces generated through passive self-ligation result in less periodontal ischemia and therefore minimal discomfort. However, in view of the low study quality of included trials, these results should be viewed with caution. Methods: At baseline, into treatment, at end of active treatment and at 7-year follow-up, the patients will be asked to answer validated questionnaires suitable for their age group about pain in the jaws and face.

Expected outcome: In the initial phase of treatment, patients will experience less pain with the new technique compared to the conventional technique. This is related to lower resistance in friction and less force needed to produce tooth movement.

Specific aim 6:To evaluate self-perceived oral health-related quality of life (OHRQoL) and working alliance formation Rationale: Few studies were identified on patient perception after orthodontic treatment, and only one of these fulfilled the criteria of a 5-year follow-up. Conclusions on patient perception in the long term were not possible to draw. For other oral conditions caregivers seem to overestimate the burden of dental conditions as compared to the patients. We find it motivated to analyze the perception of a young age-group. Methods: At baseline, into treatment, at end of active treatment and at 7-year follow-up, the patients will fill out validated questionnaires of OHRQoL. One is the EQ-5D-Y, a standardized instrument for use as a measure of health outcome in children and adolescence (1990 EuroQol Group©). The other instrument is the Children Perception Questionnaire (CPQ 11-14) Workingalliance formation will be assessed using the Working Alliance Inventory - Short Revised form (WAI-SR).

Expected outcome: Among the patients with relapse, the OHRQoL will be affected. This will be related to factors of treatment as well as the working alliance formation. The null-hypothesis is that the impact of gender will be of no significance when evaluating quality of lifevariables. Key action 4 - Evaluating treatment outcomes on a societal level Specific aim 7: To perform a cost-effectiveness analysis Rationale: Economic evaluations of methods are important and relevant for decision-making in order to allocate resources. No prospective cost-effectiveness analysis has been performed for orthodontic treatment.

Method: The total costs as well as the distribution of costs will be calculated from different perspectives. Various outcomes measures will be used (such as number of successful treatments and pain measured on a visual analogue scale), but we will also estimate quality-adjusted life-year (QALY) weights of the health states related to the two techniques. QALY weights will be created using both indirect methods (such as the EQ-5D-Y) and direct methods (such as the visual analogue scale). Using this method, the incremental cost-effectiveness ratio of self-ligating brackets can be analyzed and compared with the costeffectiveness of many other treatments. Expected outcome: The system with self-ligating brackets is more expensive to purchase. As less chair-side time is needed it will give lower total costs. The outcomes are expected to be improved with the self-ligating brackets but the scales of these effects are unknown. The cost-effectiveness is therefore unclear, but if outcomes are improved at lower cost, the self-ligating brackets will prove to be dominant.

ELIGIBILITY:
The eligibility criteria were set as follows:

* Age at treatment start: 12-17 years
* Crowding and displaced teeth
* Maximum one cusp width deviation from normal sagittal relation
* Overbite ≥ 0 mm
* Normal or only dentoalveolar transversal discrepancy
* No missing permanent teeth up to first molars
* Treatment needed according to IOTN or ICON index and treated in accordance with the Swedish system of free child and youth dental care

The exclusion criteria were set as:

* Skeletal anomalies
* Rheumatoid arthritis
* Previous orthodontic treatment
* Impacted teeth
* Ongoing sucking habits
* Previous trauma to teeth or jaws with subjective, clinical, or radiographic signs: periapical pathology; probing depth ≥ 5 mm at ≥ 4 surfaces of central incisors or first molars
* Visible plaque grade 3
* Treatment plan including extractions or other appliances than fixed buccal appliances
* Communication difficulties.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 131 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluating change in treatment outcomes at the clinical level | 2 years
  The patients will be documented with dental casts at baseline, after 9-12 months treatment and at end of active treatment. To evaluate change in tooth alignment, function stability and treatment success Peer Assessment Rating index (PAR) will be used on dental casts. PAR scores are assigned to different malocclusion traits and the difference between pre- and posttreatment scores indicates the degree of improvement as a result of orthodontic intervention.
Evaluating longitudinal change in treatment outcomes | 5 years
  The patients will be documented with dental casts end of active treatment and 5 years after active treatment. To evaluate change in stability Peer Assessment Rating index (PAR) will be used on dental casts.

SECONDARY OUTCOMES:
To evaluate the rate of root resorption and marginal bone loss after treatment | 2 years
  Clinical and radiographic examinations will be performed at baseline, after 9-12 months, at end of active treatment. (2 yrs). Intraoral radiography and CBCT will be performed to examine and measure the the tooth roots and supporting bone tissue (mm). Measuring methods with high reliability will be used
To evaluate caries incidence | 2 years
  Clinical examination, bitewing radiographs and intraoral photographs will be performed at baseline, at end of active (2yrs) treatment to examine the incidence of initial and manifest carious lesions at all tooth surfaces with validated index.
To assess pain experienced by the patients with a validated Visual Analog Scale | 2 years
  At baseline, into treatment, at end of active treatment, the patients will be asked to answer validated Visual Analog scale for pain.
  validated questionnaires suitable for their age group about pain in the jaws and face
To perform a cost-effectiveness analysis | 2 years
  The total costs as well as the distribution of costs will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Liselotte Paulsson, Study Chair — Malmö University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matilainen LB, Johansson K, Wiaderny M, Brechter A, Petren S, D'Anto V, Paulsson L. Treatment Effects and Treatment Time in Adolescents With Crowded and Displaced Teeth Treated With Fixed Appliance Systems Without Extractions: A Multi-Centre Randomised Controlled Trial. Orthod Craniofac Res. 2025 Dec;28(6):929-942. doi: 10.1111/ocr.70005. Epub 2025 Jul 23. PMID 40698883
- [Derived] Johansson K, Christell H, Brechter A, Paulsson L. Evaluation of External Apical Root Resorption and the Relevance of Intermediate Radiography in Non-Extraction Treatment With Fixed Appliances for Adolescents With Crowding: A Multicenter Randomised Controlled Trial Using CBCT. Orthod Craniofac Res. 2025 Jun;28(3):515-526. doi: 10.1111/ocr.12903. Epub 2025 Feb 3. PMID 39899339